CLINICAL TRIAL: NCT03513081
Title: Children Food Neophobia - a Playful Intervention at a Kindergarten
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Politécnico de Leiria (Other)
Collaborators: Universidade do Porto (Other)
Responsible Party: Principal Investigator, Cátia Braga-Pontes, Clinical Investigator, Instituto Politécnico de Leiria
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ChildNeophobia
Record Dates: First submitted 2018-04-16; First posted 2018-05-01 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Preschool Children
Keywords: food neophobia; preschool; children
MeSH Terms: conditions — Avoidant Restrictive Food Intake Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educative Session (Experimental): The experimental group receive nine educational sessions (one per week) about different vegetables and, at lunch time, they are exposed to a different vegetable. If they try it, they will receive a sticker. In each session, researcher will record their preference for the vegetable and the quantity that they consumed in a scale from one to three (1- the child tasted it; 2 - the child repeated it; 3 - the child ate all the quantity). In the end of 9 sessions, all children (experimental and control group) will receive the same salad that they had eaten at baseline and the procedure will be the same: the salad is weighted before and after the consumption of each child to verify the quantity of each one ate.
  Interventions: Behavioral: Educative session
- Control (No Intervention): Children in the control group don´t receive an educative session. Before the study starts children are asked to eat a salad. After 9 weeks, all children in the control group will receive the same salad that they had eaten at baseline and the procedure will be the same: the salad is weighted before and after the consumption of each child to verify the quantity of each one ate.

INTERVENTIONS:
Behavioral: Educative session — The experimental group receive nine educational sessions (one per week) about different vegetables and, at lunch time, they are exposed to a different vegetable. If they try it, they will receive a sticker. In each session, researcher will record their preference for the vegetable and the quantity that they consumed in a scale from one to three (1- the child prooved it; 2 - the child repeated it; 3 - the child ate all the quantity). In the end of 9 sessions, all children (experimental and control group) will receive the same salad that they had eaten at baseline and the procedure will be the same: the salad is weighted before and after the consumption of each child to verify the quantity of each one ate.
  Arms: Educative Session

SUMMARY:
The aim of this project is to investigate the efficacy of taste exposure-plus small reward in acceptance and consumption of vegetables among preschool children at school. In this context, interventions were attended at school in order to capture the influence of this environments towards consumption of vegetables among preschool children. For this, the methodology applied will be a repeated exposure protocol by introducing small rewards to encourage children to taste an unfamiliar or dislike food. Child intake (weight or number of pieces) and liking (hedonic scale) will be assessed at baseline sessions and exposure sessions. Moreover, child's neophobia will be evaluated and additional determinants of child neophobia, such as child's eating behaviour

DETAILED DESCRIPTION:
Food neophobia, understood as the rejection of novel foods, is considered one of the biggest barriers to the consumption of fruits and vegetables in preschool children. Some factors like food preferences, gender, genetic characteristics, psychological factors and family factors are also crucial for the acceptance of vegetable in childhood. Some strategies used to modify food preferences of children are repeated exposure and the use of rewards. The aim of this project is to investigate the efficacy of taste exposure-plus small reward in acceptance and consumption of vegetables among preschool children at school. In this context, interventions were attended at school to capture the influence of this environment towards consumption of vegetables among preschool children.

For this, the methodology applied will be a repeated exposure protocol by introducing small rewards to encourage children to taste an unfamiliar or dislike food. Child intake (weight or number of pieces) and liking (hedonic scale) will be assessed at baseline sessions and exposure sessions. Moreover, child's neophobia will be evaluated and additional determinants of child neophobia, such as child's eating behaviour. Quantitative data analysis will be performed by software IBM-SPSS Statistics®. In conducting this research is expected to achieve techniques to overcome neophobia in preschool children and promote vegetable consumption in school and at home. The results may contribute to improve food quality in childhood and consequently in adulthood.

ELIGIBILITY:
Inclusion Criteria:

* children attending an educational institution

Exclusion Criteria:

* children with cognitive impairment

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 82 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2016-02-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Child Food Neophobia | 4 months
  Child Food Neophobia Scale (Pliner 1994) - this scale is composed of ten questions, being answered by parents in a scale from one to seven, in which number one means "very similar to the reality of my child" and seven means "extremely distant to the reality of my child". This scale is able to evaluate child's food neophobia and child's food neophilia
Child Eating Behaviour | 4 months
  Child Eating Behaviour Questionnaire (Wardle, Guthrie et al. 2001) translated and adapted for portuguese reality by Viana et al (Viana and Sinde 2008). This questionnaire is answered by parents to evaluate child's eating behaviour and is composed of 35 questions. In each question the answer is in a scale from one to five, in which one means "never" and five means "always".

SECONDARY OUTCOMES:
Intake of an unfamiliar salad | 4 months
  Assessing intake of an unfamiliar salad served at lunch at three distinct moments: baseline (T0), immediately following intervention with the experimental group (T1) and ten weeks after (T2) (immediately following the intervention with the control group). This third evaluation will allow measuring the impact of the intervention at a longer period of time (Laureati, Bergamaschi et al. 2014)

CONTACTS AND LOCATIONS:
Overall Officials: Luis Cunha, PhD, Principal Investigator — Universidade do Porto

IPD SHARING:
Plan to Share IPD: Undecided